CLINICAL TRIAL: NCT04131309
Title: Phase 2 Study of Daratumumab Monotherapy in Previously Untreated Patients With Stage 3B Light Chain (AL) Amyloidosis
Brief Title: A Study of Daratumumab Monotherapy in Previously Untreated Patients With Stage 3B Light Chain (AL) Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting European Myeloma Network (Network)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Organization: European Myeloma Network B.V. (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMN22/54767414AMY2005; 2018-004333-33 (EudraCT Number)
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Light Chain (AL) Amyloidosis, Stage 3B
MeSH Terms: conditions — Amyloidosis | interventions — daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab (Experimental): Daratumumab monotherapy 16 mg/kg intravenous infusion (iv) or 1800 mg subcutaneous injection (sc) weekly for Cycles 1-2, every 2 weeks for Cycles 3-6 and every 4 weeks thereafter.
  Subjects who do not achieve either a hematologic VGPR or better, OR a hematologic PR with a major organ response by Cycle 4 Day 1 may receive, in addition to daratumumab, bortezomib (for a maximum of 6 cycles) and low dose dexamethasone.
  Interventions: Drug: Daratumumab; Drug: Bortezomib Injection; Drug: Dexamethasone oral tablet

INTERVENTIONS:
Drug: Daratumumab — As of Protocol Amendment 1, all new subjects are dosed with daratumumab subcutaneous injection (SC) co-formulated with recombinant human hyaluronidase rHuPH20. Subjects who already began treatment with daratumumab intravenous (IV) infusion (i.e., prior to Am 1) switch to SC on the next administration date according to the protocol schedule. Subjects receive daratumumab IV at a dose of 16 mg/kg and daratumumab SC at a fixed dose of 1800 mg for the first 8 weeks (Cycles 1 and 2) of treatment and then every 2 weeks for 4 cycles (Cycles 3 to 6) and then every 4 weeks until progression of disease (according to MOD-PFS), unacceptable toxicity or subsequent therapy, for a maximum of 2 years in total. All treatment cycles are 4 weeks (28 days) in length.
Drug: Bortezomib Injection — Subjects who do not achieve either a hematologic VGPR or better, OR a hematologic PR with a major organ response by Cycle 4 Day 1 may receive at Investigator's discretion, in addition to daratumumab, bortezomib at a dose of 1.3 mg/m2 weekly for a maximum of 6 cycles as a subcutaneous injection
  Other Names: velcade
Drug: Dexamethasone oral tablet — Subjects who do not achieve either a hematologic VGPR or better, OR a hematologic PR with a major organ response by Cycle 4 Day 1 may receive at Investigator's discretion, in addition to daratumumab low dose dexamethasone at a maximum total dose of 20 mg weekly.

SUMMARY:
This is an open-label, multicenter, Phase 2 study in subjects with newly diagnosed stage 3B light chain (AL) amyloidosis.

DETAILED DESCRIPTION:
The current study aims to investigate daratumumab as a monotherapy in patients with stage 3B AL amyloidosis who have not received prior therapy. Approximately 40 subjects will receive primary therapy with daratumumab. Subject participation will include a Screening Phase, a Treatment Phase, a Post-Treatment Observation Phase, and a Long-term Follow-up Phase.

A safety run-in will be conducted in 6 subjects treated with daratumumab for at least 1 cycle to establish safety of daratumumab in patients with stage 3B AL amyloidosis. Dosing of these 6 subjects will be staggered so that no subject will receive their first dose sooner than 48 hours after the previously enrolled subject. Safety evaluation will be performed by a Data Safety Monitoring Board (DSMB) after at least 1 cycle is completed for all 6 subjects. If no safety signal is observed, the enrollment of the rest of the patients will begin.

In Protocol Version 1.0, subjects receive daratumumab IV at a dose of 16 mg/kg. As of Protocol Amendment 1, all new subjects are dosed subcutaneously with daratumumab co-formulated with recombinant human hyaluronidase rHuPH20 (daratumumab SC). Subjects who already began treatment with daratumumab IV (i.e., prior to Amendment 1) switch to daratumumab SC on the next administration date according to the protocol schedule. Subjects receive daratumumab IV at a dose of 16 mg/kg and daratumumab SC at a fixed dose of 1800 mg for the first 8 weeks (Cycles 1 and 2) of treatment and then every 2 weeks for 4 cycles (Cycles 3 to 6) and then every 4 weeks until progression of disease (according to MOD-PFS), unacceptable toxicity or subsequent therapy, for a maximum of 2 years in total. All treatment cycles are 4 weeks (28 days) in length.

Subjects who will not achieve either a hematologic VGPR or better, OR a hematologic PR with a major organ response by Cycle 4 Day 1 may receive at Investigator's discretion, in addition to daratumumab, bortezomib (1.3 mg/m2 weekly for a maximum of 6 cycles) and low dose dexamethasone (total maximum weekly dose of 20mg).

ELIGIBILITY:
Inclusion Criteria:

* KEY INCLUSION CRITERIA

  1. Men or women 18 years of age or older.
  2. Diagnosis of amyloidosis, AL type, based on:

     1. Histopathological diagnosis of amyloidosis based on detection by immunohistochemistry and polarizing light microscopy of green bi-refringent material in Congo Red stained tissue specimens (excluding bone marrow) or characteristic electron microscopy appearance

        Considerations for specific populations where other types of amyloidosis may be encountered:

        • For male subjects over 70 years of age who have cardiac involvement only, and subjects of African descent (black subjects), mass spectrometry, immunoelectron microscopy, or other immunohistochemistry-based typing of AL amyloid in a tissue biopsy or a negative bone scintigraphy with Tc99m-PYP or -DPD is recommended to rule out other types of amyloidosis such as age related amyloidosis and/or hereditary amyloidosis (ATTR mutation) AND
     2. Measurable disease of amyloid light chain amyloidosis as defined by at least ONE of the following:

        * serum monoclonal protein ≥0.5 g/dL by protein electrophoresis (routine serum protein electrophoresis and immunofixation performed at local lab),
        * serum free light chain (FLC) ≥2.0 mg/dL (20 mg/L) with an abnormal kappa:lambda ratio or the difference between involved and uninvolved free light chains (dFLC) ≥2mg/dL (20 mg/L). Serum free light chains (FLCs) will be measured using the Freelite assay at a central laboratory
        * Note: Measurable disease by Urine Bence-Jones Proteinuria is not sufficient for study enrolment.

        AND
     3. Cardiac involvement by AL amyloidosis according to consensus guidelines
  3. Mayo Stage 3B disease, defined as both A. increased cardiac troponin (hsTnT > 54 pg/ml) AND B. increased NT-proBNP ≥ 8500 pg/ml
  4. For subjects with congestive heart failure, symptoms should be optimally managed and clinically stable with no cardiovascular-related hospitalizations within 2 weeks prior to Cycle 1 Day 1, as assessed by the Principal Investigator. [See also exclusion criteria 3]
  5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1, 2 or 3
  6. Subject must have pre-treatment clinical laboratory values meeting the following criteria during the Screening Phase:

     1. Absolute neutrophil count ≥1.0 × 109/L;
     2. Hemoglobin level ≥8.0 g/dL (≥5 mmol/L)
     3. Platelet count ≥75 × 109/L; platelet transfusions are NOT acceptable
     4. Alanine aminotransferase level (ALT) ≤2.5 x the upper limit of normal (ULN);
     5. Aspartate aminotransferase (AST) ≤2.5 x ULN
     6. Total bilirubin level ≤1.5 × ULN, except for subjects with history of Gilbert Syndrome, in which case direct bilirubin ≤ 2 × ULN
     7. Estimated Glomerular Filtration Rate (eGFR) ≥20 mL/min; Please note that the eGFR is measured using the CKD-EPI equation
  7. Women of childbearing potential must commit to either abstain continuously from heterosexual sexual intercourse (if this is the preferred and usual lifestyle of the subject) or to use 2 methods of reliable birth control simultaneously. This includes one highly effective form of contraception (tubal ligation, intrauterine device, hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin prior to dosing and continue for 1 year after discontinuation of cyclophosphamide or 3 months after discontinuation of daratumumab, whichever is longer. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy or bilateral oophorectomy.
  8. During the study and for 3 months after receiving the last dose of daratumumab, female subjects must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction.
  9. A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control, e.g. either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository during and up to 3 months after discontinuation of daratumumab. All men must not donate sperm during the study and for 3 months after discontinuation of daratumumab.
  10. Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to Cycle 1 Day 1. For requirements during the Treatment Phase, please see the Time and Events Schedule.
  11. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of the procedures required for the study and are willing to participate in the study. Subjects must be willing and able to adhere to the prohibitions and restrictions specified in this protocol, as referenced in the ICF.

Exclusion Criteria:

Any potential subject who meets any of the following criteria will be excluded from participating in the study:

1. Prior therapy for AL amyloidosis or multiple myeloma with the exception of 160 mg dexamethasone (or equivalent steroid) prior to Cycle 1 Day 1
2. Previous or current diagnosis of symptomatic multiple myeloma including the presence of lytic bone disease, plasmacytomas, ≥ 60% plasma cells in the bone marrow, and/or hypercalcemia.
3. Evidence of significant cardiovascular conditions as specified below:

   1. New York Heart Association (NYHA) classification of heart failure, stages IIIB or IV
   2. Heart failure that in the opinion of the investigator is on the basis of ischemic heart disease (eg prior myocardial infarction with documented history of cardiac enzyme elevation and electrocardiogram (ECG) changes) or uncorrected valvular disease, and not due to AL amyloid cardiomyopathy
   3. Hospitalization for unstable angina or myocardial infarction, or percutaneous cardiac intervention with recent stent, or coronary artery bypass grafting, all within 6 months prior to first dose
   4. Subjects with a history of sustained ventricular tachycardia or aborted ventricular fibrillation or with a history of atrioventricular (AV) nodal or sinoatrial (SA) nodal dysfunction for which a pacemaker/ICD is indicated but will not be placed (subjects who do have a pacemaker/ ICD are allowed in the study)
   5. Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >500 msec. Subjects who have pacemaker may be included regardless of calculated QTc interval.
   6. Supine systolic blood pressure <90 mmHg, or symptomatic orthostatic hypotension, defined as a decrease in systolic blood pressure upon standing of >20 mmHg despite medical management (e.g. midodrine, fludrocortisones) in the absence of volume depletion
4. Subjects planning to undergo a stem cell transplant during the first 6 cycles of protocol therapy are excluded. Stem cell collection during the first 6 cycles of protocol therapy is permitted
5. Diagnosed or treated for malignancy other than AL, except:

   1. Malignancy treated with curative intent and with no known active disease present for ≥24 months before Cycle 1 Day 1
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   3. Adequately treated carcinoma in situ (e.g. cervical, breast) with no evidence of disease
6. Subject has known chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for subjects suspected of having COPD and subjects must be excluded if FEV1 <50% of predicted normal.
7. Subject has known moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification. (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study).
8. Subject is known to be seropositive for human immunodeficiency virus (HIV). HIV positive subjects who are stable on highly active antiretroviral therapy (HAART) with no opportunistic infections within the last 6 months are eligible.
9. Subjects known to be:

   1. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [antiHBc] and/or antibodies to hepatitis B surface antigen [antiHBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (antiHBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
   2. Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
10. Subject has any concurrent medical condition or disease (eg, active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
11. Any form of non-AL amyloidosis including, wild type or mutated (ATTR) amyloidosis.
12. Subject has known allergies, hypersensitivity or intolerance to monoclonal antibodies or human proteins, or their excipients (refer to Investigator Brochure), or known sensitivity to mammalian-derived products.
13. Subject is known or suspected of not being able to comply with the study protocol (eg, because of alcoholism, drug dependency, or psychological disorder) or the subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise their well-being) or that could prevent, limit or confound the protocol-specified assessments.
14. Subject is a female who is pregnant or breast-feeding or planning to become pregnant while enrolled in this study or within 3 months following discontinuation of daratumumab.
15. Subject has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks prior to Cycle 1, Day 1.
16. Subject has had major surgery within 2 weeks prior to Cycle 1, Day 1, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study or within 2 weeks after the last dose of study drug administration. Note: subjects with planned surgical procedures to be conducted under local anesthesia may participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
overall survival | 6 months
  To evaluate the overall survival rate at 6 months following treatment with daratumumab in frontline AL patients with stage 3B disease.

SECONDARY OUTCOMES:
overall Response Rate (ORR) | at 3 and 6 months
  ORR, rate of very good partial (VGPR) and complete (CR) hematologic response
Major Organ Deterioration Progression-Free Survival (MOD-PFS). | every 28 days from start of study treatment (cycle 1 Day1) to death or major organ deterioration 2 years with an average of 6 month
  Major Organ Deterioration Progression-Free Survival (MOD-PFS) is a composite endpoint of clinically observable endpoints and will be defined from the start of study treatment (Cycle 1 Day 1) to any one of the following events (whichever occurs first)
  • Death or Major organ deterioration
Progression Free Survival | from registration to the date of disease progression or death with a maximum of 2 years
  documentation of hematologic disease progression, or organ (cardiac, renal, or liver) progression/need for transplant, or need for additional therapy (excluding the addition of bortezomib under protocol) or death due to any cause, whichever occurs first according to central laboratory results and judged by international consensus guidelines
organ response rate (OrRR) | from registration to the date of disease progression or death with a maximum of 2 years
  Heart, Kidney, Liver
Time to hematologic response | 2 years
  to evaluate the time to response
proportion of additional treatment | every 28 days, from start of study treatment (cycle 1 Day1) until end of treatment with a maximum of 2 years, average of 6 months
  o describe the proportion of subjects who received additional treatment with bortezomib and low dose dexamethasone (at the investigator's discretion).
EORTC QLQ-C30 scores will be summarized at each time point. The relationship between response and change in domain scores will be explored. the results will also be presented in two groups (SC and IV daratumumab administration). | on day 1 of cycle 1-6 (each cycle is 28 days), every 8 weeks thereafter until end of treatment with a maximum of 2 years
  The EORTC QLQ-C30 is a 30-item questionnaire containing both single and multi-item measures. These include five functional scales (Physical, Role, Cognitive, Emotional, and Social Functioning), three symptom scales (Fatigue, Pain, and Nausea/Vomiting), a Global Health Status/ Quality-of-Life (QoL) scale, and six single items (Constipation, Diarrhea, Insomnia, Dyspnea, Appetite Loss, and Financial Difficulties). The scores ranges from 0-100, a high score for functional scales and for Global Health Status/QoL represent better functioning ability or Health-Related Quality-of-Life (HRQoL), whereas a high score for symptom scales and single items represents significant symptomatology.

CONTACTS AND LOCATIONS:
Locations (5):
- France (2):
  - Hopitaux Universitaires Henri-Mondor, Créteil
  - Hopital De Rangueil CHU, Toulouse
- National and Kapodistrian University of Athens, School of Medicine, Athens, Greece
- University Hospital San Matteo, Pavia, Italy
- UMCU, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website of the European Myeloma Network — http://ww.myeloma-europe.org/